CLINICAL TRIAL: NCT05299736
Title: Multi-Agency Study on Human Impact Exposure Onboard High-Speed Boats
Brief Title: Human Impact Exposure Onboard High-Speed Boats
Acronym: MASHIEN
Status: Enrolling by invitation | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: University of Chichester (Other); Institute of Aviation Medicine, Oslo, Norway (Other Government); Naval Health Research Center (U.S. Federal Agency); German Naval Institute of Maritime Medicine / Schifffahrtmedizinisches Institut der Marine (Unknown); Fraunhofer Institute for Interfacial Engineering and Biotechnology (Other)
Responsible Party: Sponsor
Other Study IDs: MASHIEN; NATO STO HFM RTG 344 (Other: NATO STO)
Record Dates: First submitted 2022-02-21; First posted 2022-03-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Injuries; Traumatic Injury of Spine; Traumatic Head Injury
MeSH Terms: conditions — Wounds and Injuries; Spinal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Operating high-speed boats is dangerous. The purpose of this study is to establish what levels and what characteristics of impact exposure cause injuries.

Impact-induced injuries are sometimes severe and cause permanent disabilities. The slamming-impact exposure causes more injuries per workday than seen in most other peacetime work. 12.

It is however NOT known which levels or kinds of impacts are dangerous and which are safe or sustainable. To prevent injuries and to reduce fatigue onboard high-speed boats, this knowledge is crucial.

Current standards and regulations lack relevance. They are based on mean values of vibrations, and the stated exposure limit values are impossible to comply with even in normal maritime operations.

The purpose of this study is to establish what levels and what characteristics of impact exposure cause injuries.

This prospective observation study will measure human impact exposure and correlate this to the occurrence and development of pain, used to indicate the risk of injury.

DETAILED DESCRIPTION:
INTRODUCTION The ultimate purpose of the study is to protect professionals operating high-speed boats from severe impact-induced injuries.

This requires establishing what kinds of impacts are dangerous and defining relevant limits for sustainable human impact exposure.

Human impact exposure onboard high-speed boats causes pain and injuries, some severe, permanent, and debilitating, physical fatigue, and cognitive impairment.

Increasing speeds and increasing numbers of high-speed boats used in professional operations seem to increase these problems both in numbers and severity worldwide.

A lack of knowledge about the actual exposure and understanding of the causes of injuries, and the implementation of counterproductive regulations, test methods, specifications may have contributed to the increasing number of injuries.

To determine what impact exposure is dangerous, it is necessary to conduct a prospective longitudinal study on humans being subjected to the relevant actual real-life exposure at sea and correlate this exposure in real-time to a physiologic parameter indicating the risk of acute injury.

Based on the new knowledge, relevant exposure limits can be proposed to protect operators from injury and allow full operational capability underway and at target or mission.

The new facts may also lay the basis for a new quantitative measurement unit representing the impact-induced forces challenging the anatomical structures and based on the magnitude and characteristics of the impacts.

2. BACKGROUND A recent retrospective web survey of self-reported injuries on retired US SOF (Special Operations Forces) HS boat operators, the SWCC2020 survey, indicates a significant increase in injuries compared to a similar survey done on active duty personnel 20 years earlier, Ensign 2000.

The SWCC shows 1.1 injury per person per year served, 50% of injuries affecting the spine, 33% of respondents having been unconscious onboard due to whole-body impacts, 40% of respondents have a VA Disability rating of 70 to 100%.

This is an extreme work environment, and relatively few individuals in each country are exposed. Hence, there are still significant knowledge gaps that must be filled to solve the problems:

What is the actual exposure? When does it get dangerous? Which impact characteristics do affect the risk of injury? How should these characteristics be weighed against each other? As the impact exposure is unpredictable and stochastic, it is impossible to simulate in an artificial environment.

The human body is a highly intricate "apparatus" designed to protect itself from noxious exposure in several ways: It is also extremely difficult to predict the physiological response from an unlimited variety of impacts. The body has 360 joints, 206 bones, and 600 muscles reacting to sudden external forces.

Many physiological factors influence how impacts affect the human body: bodyweight, stature, central gravity, posture, muscular strength, physical shape, training status of the reflex response, etc.

Many physical factors influence how impacts affect the human body: various characteristics of the impacts such as peak acceleration value, rise time, frequency content, impact duration, impact period, number of impacts, the direction of impact/force vectors, etc.

The lack of relevant knowledge has led to non-relevant exposure regulations based on non-relevant measurement standards. The EU directive 2002/44, designed to control occupational exposure to continuous vibration, is based on the ISO vibration standard 2631. These documents use VDV, Vibration Dose Value, to quantify exposure to continuous vibration. VDV has been shown to lack correlation to exposure to severe discrete impacts. Sed(8) has been suggested but is also designed to quantify continuous vibration and has the same limitations.

The vibration exposure limits stipulated by the EU directive 2002/44 lacks relevance for exposure to discrete impacts. These limits are also impossible to comply with while conducting sea rescue, law-enforcement missions, or military training in normal sea conditions.

Hence, they are disregarded in most nations, and operators lack relevant regulatory protection.

This study is based on the following facts: F. and assumptions: A. F. Hull impacts at sea can exceed 20 g peak value. A. Higher peak values cause higher risks of injuries. F. Rise times (time from 0 to peak g) of impacts can be as short as 6 ms A. Shorter rise times can cause higher and more dangerous impulses. F. Impacts containing lateral forces cause more injuries than purely vertical A. Impact exposure must be measured so that three force vectors, x,y, and z, can be analyzed.

F. Impacts measured on a seat differ significantly from impacts measured on humans.

A. Impact exposure measured on the human is more relevant than exposure measured on the seat.

F. Horizontal impacts forces on humans cannot be measured on a seat. A. Human impact exposure must be measured on the human body. F. Low pass filtering of impact data hides the information about peak values and rise times A. Exposure data must be collected as unfiltered raw data. F. Converting exposure data into VDV or Sed(8) changes peak values and rise times.

A. Exposure data must be collected as raw, unfiltered data. F. Pain can exist without injury, but acute injury normally causes pain. F. Pain can be scientifically monitored using the Nordic Minister Council PainDrawing form.

A. Events and persistence of pain can be used to indicate incipient injury.

3. METHOD The purpose of the study is to correlate impact exposure on boat hulls and humans to a physiological parameter possible to use as an indicator of developing an injury. The only such parameter possible to monitor daily in a cohort of hundreds is pain.

As this non-intervention study aimed to establish the actual normal exposure, exposure data will be collected only during normal regular activities, and no transits will be done for the purpose of collecting data.

The research method is designed to record impact exposure on hulls and humans onboard boats operating in real sea conditions. Accelerations will be recorded as unfiltered, raw data. This will allow for analysis of all the characteristics of impacts, potentially relevant for physiological effects and risks of injury. This shall make it possible to assess the significance of not only peak acceleration values but also of rise-times (time from 0 g to peak g), impact duration, energy content, slam period (time between slams), and force vector (direction of impact), etc. This will also make the results transparent and possible to scrutinize.

3.1 MULTI-AGENCY STUDY DESIGN The collaborative effort aims to gather sufficient volumes of data to reach statistical power. This requires all agencies to use the same study protocols, hardware, and software and eventually share the relevant results in a shared database.

Agencies in 16 nations have already expressed their interest in participating. All subject data will be anonymous and boat data stripped of potentially sensitive operational information before being submitted to the shared database.

Crucial synergies can also be achieved by sharing costs, data, and results. To achieve statistically significant results, a sufficient number of boats, subjects, and wave-slam events can be gathered.

3.2 MEASURING IMPACTS ON HUMANS AND HULLS Whole-body impact will be monitored on two people on board each boat at all times. Each boat will have a data logger installed for the entire study period. This will be connected to a 3-axis accelerometer attached to the hull, close to its COG. Two crew, preferably the coxswain and navigator, will wear 3-axis accelerometers mounted to kidney belts and connected to the data logger. Recorded data will indicate the actual, real-life impact exposure and the forces acting on the hulls and humans. This data will show the real exposure and the relation between hull impacts and human impacts for each boat type.

3.3 DATA LOGGER AND SENSORS A bespoke data logger device has been developed for this study. MAREC (Marine Acceleration Recorder) is optimized for ease of use and installation. Installed onboard and connected to 12 or 24 V DC, it will automatically start recording as soon as the boat makes a speed of more than 3 kts. MAREC has 10 analog channels, of which 9 are used for the three 3-axis accelerometers with a ± 25 g range. The sampling rate will be 600Hz. It also has a built-in GPS receiver logging satellite time, position, heading, and speed. The 16 Gb internal USB memory can store the data for the entire period of the study. Afterward or even during the study, the data can be uploaded to a PC for analysis.

3.4 PAIN INDICATES RISK OF INJURY Pain is used to indicate if exposure causes a risk of injury. All personnel serving onboard the boats will log events and development of pain during the entire trial period.

A bespoke smartphone app, PainDrawing, will prompt subjects daily to log any relevant pain. This is built on two scientifically validated methods, VAS, Visual Analogue Scale, and the Nordic Ministers Council's pain-drawing form. The app can be downloaded for free for both Android and iPhone.

Pain is the only physiologic parameter that can be used as an indicator of risk of injury and be monitored and quantified over time, frequently enough to monitor a large cohort. Its function is to prevent injury. Pain can be present without injury, but rarely an acute injury manifests without pain.

Pain is also a relevant symptom, or sometimes a condition, which compromises physical performance, endurance, and even mental capacity. It should be evident that exposure causing pain during demanding operations must be avoided or limited as much as possible.

3.5 DATA ANALYSIS AND MANAGEMENT Participating agencies and organizations will upload the collected exposure data to their local computers. The binary files will be converted and presented in a graphic format legible even by laypersons.

The data analysis software will then select the relevant non-sensitive part for sharing and, on command, be uploaded to a common big-data database.

A data analysis engine DAE, built for the purpose, will analyze the correlation of the various characteristics of the impacts to the physiological response, reported as experience and persistence of pain.

4. RESULTS AND APPLICATIONS Based on the expected results of the study, it will be possible to calibrate instruments with dashboard-mounted indicators, telling operators when hull impacts exceed safe levels by green, yellow, or red signals, where red should indicate out of boundaries.

The results should also indicate the significance of the various analyzed impact characteristics.

Ultimately the results can lay a base for relevant recommendations for allowable versus dangerous levels of exposure to whole-body impact.

Participating agencies will gather information about how their various boats perform, producing slamming impacts in actual use. They will also be able to see how various levels of operator skills affect exposure.

5. CONCLUSION Current standards and regulations cannot quantify or help control human impact exposure at sea.

In many fields of medical science, it is only possible to get relevant answers by studying the human itself. In this case, the new knowledge needed to solve the problem can only be established by studying what happens in real life.

Scientists and medical professionals have a duty to implement State-of-the-Art knowledge to find the facts needed to solve these severe occupational health problems. Hence, the investigators have chosen an empirical approach, investigating what happens to humans in real-life at sea.

ELIGIBILITY:
Inclusion Criteria:

• Volunteering crew or passengers working onboard or being transported in a professional capacity onboard boats used by the participating agencies and organizations

Exclusion Criteria:

• Nonvolunteering

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All volunteering regular crew or passengers working onboard or being transported in a professional capacity onboard boats used by the participating agencies and organizations.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak acceleration levels of actual human impact exposure onboard High-Speed boats | May 2022 - Dec 2022
  This will show the peak acceleration levels to which humans are exposed in three directions, X, Y, and Z, relative to the boat.
  Acceleration is measured in m/s2.
Safe versus unsafe levels of real-life human impact exposure onboard H-S boats | Jan 2023 - Dec 2024
  This will indicate at what human acceleration levels injuries can be expected.

SECONDARY OUTCOMES:
Range of rise-times and correlation to peak acceleration levels | Jan 2023 - Dec 2024
  Rise time (s) measured from nominal 0 g to peak acceleration
Range of jerk and correlation to peak acceleration levels | Jan 2023 - Dec 2024
  Jerk is the derivative of the acceleration over the time from 0 g to peak acceleration, Delta acc/Delta t)(m/s3)
Total mechanical effect (Watt) in impacts . | Jan 2023 - Dec 2024
  The total mechanical effect of each discreet impact can be calculated. This measure may correlate to the physiological response. Mechanical effect is measured in Watt.
Correlation of various impact characteristics to reported pain. | Jan 2023 - Dec 2024
  As all the various characteristics may affect the risk of failure of anatomical structures, each one has to be analyzed and weighed against the other, and then the results correlated to the physiological response reported pain.

OTHER OUTCOMES:
Recommendation for a new relevant way to quantify human impact exposure. | Jan 2023 - Dec 2024
  This recommendation will suggest a method of measuring impact exposure on boats and on humans. It would also suggest a way of quantifying the exposure in a unit that is correlated to the risk of impact-induced injury. This unit will contain some of analyzed characteristics, weighed in in a way that will make the unit correlate to the physiological response.
Recommendation for new relevant limits for sustainable human impact exposure. | Jan 2023 - Dec 2024
  Proposal for relevant impact exposure limits can be used by agencies, to prevent injuries, to keep personnel onboard fit for mission, to maintain operational capability, and also eventually as a basis for replacing current irrelevant rules and regulations.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Myers, Professor, Study Chair — University of Chichester, Professor of Exercise Physiology
Locations (1):
- University of Gothenburg, Institution for Clinical sciences, Department of Orthopaedics, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ullman J, Myers SD, Bretschneider KT, Kelly KR, Daniel Y, Hurpin V, Kaehler J, Kasin JI, Hveding K, Mansfield N, Masouros SD, Perl D, Wijnands N, Vallee I, Stevens V, Fraser JJ, Rolfson O, Robinson Y. MultiAgency, prospective, exploratory, non-intervention, cohort Study on Human Impact Exposure oNboard high-speed boats (MASHIEN): protocol. BMJ Open. 2025 May 2;15(5):e090993. doi: 10.1136/bmjopen-2024-090993. PMID 40316357
- [Derived] Ullman J, Hengst D, Carpenter R, Robinson Y. Does Military High-speed Boat Slamming Cause Severe Injuries and Disability? Clin Orthop Relat Res. 2022 Nov 1;480(11):2163-2173. doi: 10.1097/CORR.0000000000002420. Epub 2022 Sep 30. PMID 36190503